CLINICAL TRIAL: NCT05035576
Title: A Randomized, Adaptive Design, Proof of Concept, Single Dose Study to Evaluate Change in Viral Load After OPN-019 in Adults With COVID-19
Brief Title: A Study to Evaluate Change in Viral Load After OPN-019 in Adults With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPN-PVI-COV-1401
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400 mg OPN-019 (Active Comparator)
  Interventions: Drug: OPN-019
- Standard of Care (SOC) (No Intervention)

INTERVENTIONS:
Drug: OPN-019 — 400 mg OPN-019, 2 sprays per nostril (one dose)
  Arms: 400 mg OPN-019

SUMMARY:
The purpose of this study is to determine both the magnitude and duration of viral load (copies/mL) reduction after a single dose of OPN-019. The variability associated with viral counts will be utilized to inform the study design of future studies.

DETAILED DESCRIPTION:
A randomized, single dose, adaptive design, proof of concept study in subjects who have tested positive for SARS-CoV-2 infection, are recently infected, and who have mild or no symptoms. Patients will be required to have a score ≤ 2 on the WHO ordinal scale for clinical improvement (Covid-19 Therapeutic Trial Synopsis; Feb 18, 2020). Those meeting the inclusion criteria will be randomized to 1 of 2 arms: OPN-019 (2 sprays per nostril) or SOC. Once randomized, subjects will have baseline nasal and oropharyngeal swabs performed for qRT-PCR viral load and infectious viral particle assessment. The subject will then be administered the study medication. Subsequent nasal and oropharyngeal swabs will be taken at 1 hour, 3 hours, 6 hours, 8 hours, 12 hours, and 24 hours. Cohorts of 10 subjects will be randomized into the study and the results from those subjects will be evaluated to determine if changes in the inclusion criteria or study assessments are required.

ELIGIBILITY:
Inclusion Criteria:

1. men or women aged 18 years and older at Visit 1 (Baseline/Screening)
2. women of child-bearing potential must have a negative urine pregnancy test at Visit 1 (Baseline/Screening)
3. must be confirmed positive for SARS-CoV-2 with RT-PCR testing of a nasal swab taken within 72 hours prior to randomization (first dose of study drug)
4. must have a score ≤ 2 on the WHO ordinal scale for clinical improvement
5. subject must be willing to refrain from any other intranasal instillations (e.g., medications, saline, etc.) for 24 hours after study medication dosing
6. must be capable, in the opinion of the investigator, of providing informed consent to participate in the study.

Exclusion Criteria:

1. women who are pregnant or lactating
2. hospitalized subjects or subjects requiring nursing care for COVID-19
3. currently has one of the clinical signs suggestive of moderate-to-severe COVID-19 illness:

   1. O2 saturation of ≤ 93% on room air at sea level
   2. Heart rate ≥ 90 beats per minute (after seated for 5 min)
   3. Respiratory rate ≥ 20 breaths per minute
4. receiving respiratory support (including any form of oxygen therapy)
5. history of hypothyroidism, goiter, hyperthyroidism, thyroid tumor, autoimmune thyroid disease
6. currently taking medications that contain iodine or currently taking lithium
7. receiving any other investigational drug
8. has an allergy, hypersensitivity, or contraindication to povidone iodine
9. has an allergy or hypersensitivity to any excipients in study medication
10. any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in nasal viral load over multiple time points | Baseline, 1 Hour, 3 Hours, 6 Hours, 8 Hours, 12 Hours, 24 Hours post dosing/randomization
  Change in nasal viral load (copies/mL) over multiple time points as measured by qRT-PCR testing of nasal swabs.

SECONDARY OUTCOMES:
Cumulative viral load over 6, 8, and 12-hour periods in oropharyngeal swab | 6 Hours, 8 Hours, 12 Hours post Dosing/Randomization
  Compare cumulative viral load (copies/mL) (total) over 6, 8, and 12-hour periods in oropharyngeal swab measured by qRT-PCR
Cumulative amount of Nasal Swab infectious viral particles | Baseline, 24 Hours post dosing/randomization
  Compare cumulative amount of infectious viral particles (copies/mL) between OPN-019 dosed subjects versus SOC control group in nasal swab
Number of subjects with viral load of <10^6 copies/mL | Baseline, 24 Hours post dosing/randomization
  Compare the number of subjects who reach a viral load (copies/ml) of <10^6
Maximum log reduction in viral load | Baseline, 24 Hours post dosing/randomization
  Compare maximum log reduction in viral load (copies/ml) by qRT-PCR
Time Comparison-subject virus-free or has viral load of <10^6 copies/ml | Baseline, 24 Hours post dosing/randomization
  Time over which subject is virus-free or has viral load (copies/mL) of <10^6 , both as measured by qRT-PCR
Log viral reduction assessment in subgroups-baseline viral load | Baseline, 24 Hours post dosing/randomization
  Assess log viral reduction in subgroups by baseline viral load (copies/mL)

OTHER OUTCOMES:
Evaluation of Safety by recording the severity of spontaneously reported adverse events (AEs) | Baseline, 24 Hours post dosing/randomization
  Assessment of safety by measuring severity of spontaneously reported AEs using scale with 1=mild, 2=moderate, 3=severe
Evaluation of Safety measuring vital signs- Blood Pressure | Baseline, 24 Hours post dosing/randomization
  Includes systolic and diastolic blood pressure measurements in millimeter of mercury (mmHg)
Evaluation of Safety measuring vital signs- Pulse | Baseline, 24 Hours post dosing/randomization
  Measure pulse in beats per minute (bpm)
Evaluation of Safety measuring vital signs- Temperature | Baseline, 24 Hours post dosing/randomization
  Measure temperature in °Fahrenheit (°F)
Evaluation of Safety measuring vital signs- Respiratory Rate | Baseline, 24 Hours post dosing/randomization
  Measure Respiratory Rate in breaths per minute
Evaluation of Safety - Monitoring Concomitant Medication Usage | Baseline, 24 Hours post dosing/randomization
  Assessment for safety from the collection of information for concomitant medications usage
Evaluation of Safety - Study Drug Tolerability | 1 Hour Post Dose
  Study Medication Tolerability Questionnaire will be completed by subjects rate the levels of nasal discomfort and unpleasant taste associated with study medication use; study specific measure. The Study Medication Tolerability Questionnaire is administered verbally by a study staff member to the subject. This 11-item score is rated on a 0-100 scale, 0 being "dislike it an extreme amount", and 100 being "like it an extreme amount"

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carothers, Study Director — OptiNose US; John Messina, Study Chair — OptiNose US
Locations (1):
- Fundacion Santos y de la Garza Evia, I.B.P, Monterrey, N.L., Mexico